CLINICAL TRIAL: NCT01059604
Title: The Sumatriptan and Naratriptan Pregnancy Registry
Brief Title: Sumatriptan and Naratriptan Pregnancy Registry
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112914; EPIP082 (Other: GSK); EPI40050 (Other: GSK)
Record Dates: First submitted 2010-01-28; First posted 2010-02-01 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Migraine Disorders
Keywords: pregnancy outcomes; pregnancy; first trimester; Sumatriptan; major congenital malformations; naratriptan; sumatriptan-naproxen combination; pregnancy registry
MeSH Terms: conditions — Migraine Disorders | interventions — Sumatriptan; naratriptan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant women exposed to sumatriptan, naratriptan, or combo: Women exposed to sumatriptan, naratriptan or the sumatriptan-naproxen combination treatment during pregnancy
  Interventions: Drug: Sumatriptan; Drug: Naratriptan; Drug: Sumatriptan-naproxen combination

INTERVENTIONS:
Drug: Sumatriptan — Sumatriptan
Drug: Naratriptan — Naratriptan
Drug: Sumatriptan-naproxen combination — Sumatriptan-naproxen combination

SUMMARY:
Anti-migraine drugs, including triptans, are not indicated for use in pregnancy. However, the peak prevalence of migraine is in women of childbearing age. This, coupled with the sporadic nature of migraine attacks and high rates of unplanned pregnancies, makes unintentional exposure to anti-migraine medications during pregnancy likely. Prior to an anti-migraine medication being marketed there are few data available on drug safety in pregnancy: data from animal models may not translate directly to humans and pregnant women are routinely excluded from clinical trials. The Sumatriptan Pregnancy Registry was established by GlaxoSmithKline (GSK) in 1996 to monitor the safety of sumatriptan during pregnancy. It was combined with the Naratriptan Pregnancy Registry in 2001 and data collection on the sumatriptan-naproxen combination (Treximet) began in 2008.

DETAILED DESCRIPTION:
The Sumatriptan, Naratriptan and Treximet Pregnancy Registry aims to assess whether there is a substantial increase in the risk of major congenital malformations (MCMs) following in utero exposure to those anti-migraine medications. Exposure during the first trimester is of primary interest as this represents the period of organogenesis.

The Registry is a primarily prospective enrolment and follow-up study. Patients exposed to sumatriptan, naratriptan, or the sumatriptan-naproxen combination during pregnancy, are enrolled, on a voluntary basis, by their healthcare provider. Enrolment is encouraged early in pregnancy and if possible prior to any prenatal testing. The healthcare provider provides initial information concerning patient demographics; details of the pregnancy including the estimated delivery date and results of any prenatal testing; and the timing, dosage, route of delivery (e.g. oral, subcutaneous, intranasal) of drug exposure in pregnancy. The registry accepts exposure reports from anywhere in the world. Within the United States (US) the healthcare provider can contact the registry using a toll free number. Outside of the US enrolments are made through the GlaxoSmithKline local operating company.

Close to the estimated date of delivery the healthcare provider is contacted by the Registry to provide follow up information concerning the pregnancy outcome (live or still birth, spontaneous or induced abortion), the presence or absence of a MCM, and the history of headache and exposure to sumatriptan, naratriptan or the sumatriptan-naproxen combination during pregnancy. Up to six attempts are made to contact the healthcare provider to obtain pregnancy outcome information. After six attempts, the record is closed as lost to follow up.

Pregnancy outcomes are classified as outcomes with MCMs, outcomes without MCMs and spontaneous abortions. The outcomes with and without MCMs are further classified as live births, stillbirths/fetal deaths and induced abortions. Spontaneous abortions are reported separately due to potential for inconsistent identification of malformations in that situation.

It is beyond the scope of the Registry to consistently access pediatric evaluations and medical records. For this reason the main outcome is restricted to major congenital malformations that are external and recognizable in the delivery room or shortly after birth. To provide consistency, reported congenital malformations are classified as major or minor according to criteria used by the Centers for Disease Control and Prevention (CDC)'s Metropolitan Atlanta Congenital Defects Program (MACDP). All malformation reports are reviewed and classified by a paediatrician from the CDC and further information is requested as necessary.

Analyses are restricted to prospectively enrolled pregnancies (enrolment prior to knowledge of the birth outcome). Retrospectively enrolled pregnancies are reviewed for patterns of malformation types, but are not included in formal analyses as retrospective reporting can be biased towards more unusual and severe outcomes and are less likely to be representative of the general population experience.

The proportion of infants with MCMs among prospectively reported exposures is calculated as: the total number of outcomes with major birth defects (number of outcomes with major birth defects + the number of live births without defects).

All spontaneous pregnancy losses, as well as induced abortions and fetal deaths without reported defects, are excluded from the denominator due to the potential for inconsistent identification of malformations in those situations. The 95% confidence intervals (CIs) for risk estimates are calculated using exact methods based on the binomial distribution.

Analyses are stratified according to trimester of exposure (with the second trimester starting at week 14 and the third trimester at week 28 of gestation) for each anti-migraine of interest. If an individual is exposed to multiple drugs of interest during pregnancy, the exposure is included in analyses for each drug of interest.

The registry does not have an internal comparator group, but descriptive comparisons are made with MCM rates from general population studies in the literature.

Prospective reports are also reviewed to detect any unusual patterns of malformation types that may warrant further investigation.

The data from the Sumatriptan, Naratriptan and Treximet Pregnancy Registry are reviewed, and conclusions developed, by an independent scientific advisory committee. A semi-annual interim report summarizing aggregate data is provided to disseminate information on a regular basis.

ELIGIBILITY:
Inclusion Criteria:

* Women exposed in utero to sumatriptan, naratriptan or the sumatriptanp-naproxen combination during pregnancy. Exposure can occur at any time during pregnancy, though exposure in the first trimester is of primary interest.
* Pregnancies exposed to sumatriptan, naratriptan or the sumatriptan-naproxen combination and reported before the outcome of the pregnancy is known (prospective reporting). Ideally exposed pregnancies are registered prior to prenatal testing, but only those pregnancies enrolled after prenatal testing has diagnosed a congenital malforamtion are excluded.
* Retrospectively reported exposures (i.e. exposures registered once the pregnancy outcome is known) are included in the registry, but are considered descriptively and are not included in risk analyses.

Exclusion Criteria:

* Retrospectively reported exposures (i.e. exposures registered once the pregnancy outcome is known) are included in the registry, but are reviewed separately and descriptively. These are not included in risk analyses.
* Patient reported exposures and outcomes that are not verified by a healthcare provider.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women exposed to sumatriptan, naratriptan or the sumatriptan-naproxen combination during pregnancy anywhere in the world.
Sampling Method: Non-Probability Sample
Enrollment: 868 (Actual)
Dates: Start 2001-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Major congenital malformations (MCMs) classified according to the Centers for Disease Control and Prevention (CDC)'s Metropolitan Atlanta Congenital Defects Program (MACDP) criteria. | Although reports and diagnoses of MCMs are accepted up to six years after the birth, the majority of malformations are reported following assessments made in the delivery room or shortly after birth.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Background] Cunnington M, Ephross S, Churchill P. The safety of sumatriptan and naratriptan in pregnancy: what have we learned? Headache. 2009 Nov-Dec;49(10):1414-22. doi: 10.1111/j.1526-4610.2009.01529.x. Epub 2009 Oct 5. PMID 19804390
- [Background] Eldridge RR, Ephross SA, Heffner CR, Tennis PS, Stender DM, White AD. Monitoring pregnancy outcomes following prenatal drug exposure through prospective pregnancy registries and passive surveillance: a pharmaceutical company commitment. Prim Care Update Ob Gyns. 1998 Jul 1;5(4):190-191. doi: 10.1016/s1068-607x(98)00115-2. PMID 10838360
- [Background] Reiff-Eldridge R, Heffner CR, Ephross SA, Tennis PS, White AD, Andrews EB. Monitoring pregnancy outcomes after prenatal drug exposure through prospective pregnancy registries: a pharmaceutical company commitment. Am J Obstet Gynecol. 2000 Jan;182(1 Pt 1):159-63. doi: 10.1016/s0002-9378(00)70506-0. PMID 10649172
- [Background] Eldridge RR, Ephross SA. Monitoring birth outcomes in the Sumatriptan Pregnancy Registry. Prim Care Update Ob Gyns. 1998 Jul 1;5(4):190. doi: 10.1016/s1068-607x(98)00114-0. PMID 10838359
- [Background] Sumatriptan and Naratriptan Pregnancy Registry. Interim Report 1 January 1996 through 31 October 2009. Issued February 2010. Available at: http://pregnancyregistry.gsk.com/index.html
- See also: Click here for interim results available on the GSK Clinical Study Register — http://www.gsk-clinicalstudyregister.com/result_detail.jsp?protocolId=112914&studyId=CC0A5421-418C-413F-B0B6-12D6C0B24F03&compound=naratriptan
- See also: Click Here to See Preliminary Results on GSK's Clinical Study Register — http://www.gsk-clinicalstudyregister.com/result_detail.jsp?protocolId=112914&studyId=CC0A5421-418C-413F-B0B6-12D6C0B24F03&compound=naratriptan